CLINICAL TRIAL: NCT01823016
Title: A Phase 2a, Randomized, Double-Blind, Placebo-Controlled, Multicenter, Parallel Group Study of JNJ-38518168 in Symptomatic Adult Subjects With Uncontrolled, Persistent Asthma
Brief Title: A Study of JNJ-38518168 in Symptomatic Adult Participants With Uncontrolled, Persistent Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR100976; 38518168ASH2001 (Other: Janssen Research & Development, LLC); 2012-004920-39 (EudraCT Number)
Record Dates: First submitted 2013-03-28; First posted 2013-04-04 (Estimated); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Asthma
Keywords: Uncontrolled, persistent asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- JNJ-38518168 (Experimental)
  Interventions: Drug: JNJ-38518168

INTERVENTIONS:
Drug: Placebo — Placebo tablet, taken once daily
  Arms: Placebo
Drug: JNJ-38518168 — JNJ-38518168, 30 mg tablet, taken once daily
  Arms: JNJ-38518168

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of JNJ-38518168 compared with placebo in participants with persistent asthma that is inadequately controlled despite current treatment.

DETAILED DESCRIPTION:
This study will be randomized (treatment group assigned by chance, like flipping a coin), double-blind (study investigators and participants will not know what treatment is being administered), and placebo-controlled (a placebo is identical to the study agent, but contains no active ingredients). A total of 160 participants will receive either placebo or JNJ-38518168 once daily. The study duration will be approximately 32 weeks and will include a screening phase of approximately 4 weeks, a 24-week placebo-controlled treatment phase, and a 4-week follow-up phase. Participant safety will be monitored throughout the entire study period..

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of asthma for at least 26 weeks, confirmed by the investigator at Screening Visit 1
* Have been receiving inhaled corticosteroid (ICS) (≤1000 µg/day fluticasone or its equivalent) for at least 12 weeks prior to Screening Visit 1
* At Screening Visit 1, be receiving the same dose of ICS ≤1000 µg/day fluticasone (or equivalent) alone or in conjunction with long-acting β2-agonist (LABA) and/or montelukast for at least 4 weeks prior to screening with no changes in dose or dosing regimen of any of these therapies during that 4 week period prior to screening
* Have an Asthma Control Questionnaire (ACQ) score ≥1.5 at Screening Visit 1
* Have a prebronchodilator forced expiratory volume in 1 second (FEV1) equal to 40% to 80%, inclusive, of predicted value at Screening Visit 1
* Have a ≥12% relative change and ≥200 mL change in FEV1 postbronchodilator at either Screening Visit 1 or 2

Exclusion Criteria:

* Has ever had a life-threatening asthma attack including respiratory arrest, intubation, or intensive care unit (ICU) admission due to asthma
* Has a history of any other chronic respiratory condition including, but not limited to, chronic obstructive pulmonary disease (COPD), bronchiolitis, bronchiectasis, allergic bronchopulmonary aspergillosis (mycosis), occupational asthma, sleep apnea, pulmonary hypertension, or any other obstructive pulmonary disease
* Has any use of the following asthma therapies: systemic corticosteroids within 6 weeks of Screening Visit 1; oral beta-agonists within 4 weeks of Screening Visit 1; cromolyns within 4 weeks of Screening Visit 1; leukotriene inhibitors other than montelukast within 4 weeks of Screening Visit 1; theophylline within 4 weeks of Screening Visit 1; inhaled anti-cholinergic agents within 4 weeks of Screening Visit 1; or omalizumab within 130 days of Screening Visit 1
* Has initiated or discontinued allergen immunotherapy within 12 weeks of Screening Visit 1
* Has smoked within 3 years of Screening Visit 1 or has a history of smoking ≥ 10 pack years
* Body-Mass Index (BMI) greater than or equal to 40 kg/m2

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2013-09; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in prebronchodilator forced expiratory volume in 1 second (preBD FEV1) | Baseline to Week 16
  Expressed as percent of predicted value.

SECONDARY OUTCOMES:
Change from baseline in Asthma Control Questionnaire (ACQ) | Baseline to Week 16
  ACQ evaluates clinical impairment that participants with asthma may experience. Items are scored on a 7-point scale (0 = good control, 6 = poor control). Higher mean scores reflect poorer control.
Change from baseline in postbronchodilator forced expiratory volume in 1 second (postBD FEV1) | Baseline to Week 16
  Expressed as percent of predicted value.
Change from baseline in weekly average of daytime asthma diary symptom scores | Baseline to Week 16
  Asthma diaries include questions about the frequency/severity of symptoms and impact on activities. Higher scores indicate more asthma symptoms.
Change from baseline in weekly average of nighttime asthma diary symptom scores | Baseline to Week 16
  Asthma diaries include questions about number of nocturnal awakenings.
Change from baseline in weekly average of number of puffs in a day that rescue medication is used | Baseline to Week 16

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (54):
- United States (20):
  - Scottsdale, Arizona
  - Los Angeles, California
  - Mission Viejo, California
  - San Diego, California
  - Denver, Colorado
  - Waterbury, Connecticut
  - Minneapolis, Minnesota
  - St Louis, Missouri
  - Bellevue, Nebraska
  - Lebanon, New Hampshire
  - Rochester, New York
  - Greenville, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Medford, Oregon
  - Portland, Oregon
  - Altoona, Pennsylvania
  - Dallas, Texas
  - San Antonio, Texas
- Canada (9):
  - Calgary, Alberta
  - Vancouver, British Columbia
  - Hamilton, Ontario
  - Kingston, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Québec, Quebec
  - Sainte-Foy, Quebec
- Montpellier, France
- Germany (10):
  - Berlin
  - Frankfurt
  - Großhansdorf
  - Hanover
  - Koblenz
  - Leipzig
  - Lübeck
  - Magdeburg
  - Mainz
  - Rüdersdorf
- Israel (6):
  - Ashkelon
  - Haifa
  - Jerusalem
  - Ramat Gan
  - Rehovot
  - Tel Aviv
- United Kingdom (8):
  - Chertsey
  - Cottingham
  - Dundee
  - Glasgow
  - London
  - Portsmouth
  - Southampton
  - Wolverhampton

REFERENCES:
- [Derived] Kollmeier AP, Barnathan ES, O'Brien C, Chen B, Xia YK, Zhou B, Loza MJ, Silkoff PE, Ge M, Thurmond RL. A phase 2a study of toreforant, a histamine H4 receptor antagonist, in eosinophilic asthma. Ann Allergy Asthma Immunol. 2018 Nov;121(5):568-574. doi: 10.1016/j.anai.2018.08.001. Epub 2018 Aug 11. PMID 30102965